CLINICAL TRIAL: NCT05981508
Title: Feasibility of Conducting an Online Family Dyadic/Couple Skills Training for Black Adults Enrolled in a Behavioral Weight Loss Intervention - Together, Eating and Activity, Matter+ (TEAM+)
Brief Title: Online Family Dyadic Skills Training for Black Adults in Behavioral Weight Loss Program
Acronym: TEAM+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Splendor-NC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-1598; 5U24DK132715-03 (NIH)
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Results first posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2023-07

CONDITIONS: Body Weight; Body Weight Changes; Obesity; Overweight and Obesity; Overweight; Behavior, Eating; Physical Inactivity; Chronic Disease; Weight Loss; Weight Reduction
MeSH Terms: conditions — Body Weight; Body Weight Changes; Obesity; Overweight; Feeding Behavior; Sedentary Behavior; Chronic Disease; Weight Loss | interventions — Eating; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-person Family Skills Training (Active Comparator): The index partner will participate in intervention as a dyad with a family member with an in-person skills training.
  Interventions: Behavioral: Together, Eating and Activity, Matter Plus (TEAM+) In-Person
- Online Family Skills Training (Experimental): The index partner will participate in intervention as a dyad with a family member with an online skills training.
  Interventions: Behavioral: Together, Eating and Activity, Matter Plus (TEAM+) Online

INTERVENTIONS:
Behavioral: Together, Eating and Activity, Matter Plus (TEAM+) Online — TEAM+ is a 3-month, family enhanced behavioral weight loss (BWL) intervention designed for Black adults consisting of an online family dyadic skills training and in-person core behavioral weight loss sessions.
  Other Names: TEAM +
  Arms: Online Family Skills Training
Behavioral: Together, Eating and Activity, Matter Plus (TEAM+) In-Person — TEAM+ is a 3-month, family enhanced behavioral weight loss (BWL) intervention designed for Black adults consisting of in-person family dyadic skills training and core behavioral weight loss sessions.
  Other Names: TEAM +
  Arms: In-person Family Skills Training

SUMMARY:
The purpose of this research study is to test the feasibility and acceptability of an interactive counselor -led online family skills training as part of a behavioral weight loss program for Black Adults.

DETAILED DESCRIPTION:
Nearly half (49.9%) of Black adults in the United States live with obesity. Black adults are underrepresented in standard behavioral weight loss (BWL) interventions and experience sub-optimal weight loss outcomes when included in such programs. Cultural adaptations to BWL interventions that recognize the family behavioral context and address the cultural value of family among Black populations are needed to improve weight loss outcomes. Prior research, including our randomized controlled pilot, Together, Eating and Activity, Matter Plus (TEAM+), have incorporated family skills training to enhance family involvement, targeting cohesion and communication, in addition to core weight loss curriculum. However, family inclusion in weight loss interventions can result in additional barriers to retention and adherence.

Technology has become an attractive delivery format to increase reach to at-risk populations, as a well-designed online program can address issues of timely access and geographical location (or distance from program sites), which are linked to low retention of Black participants. However, technology uptake among Blacks populations still lags due to mistrust, skepticism, concerns about confidentiality, privacy, and remote interaction with staff. Increases in acceptance and utilization of telemedicine and mobile-health were reported during the COVID-19 pandemic. Considering the time and location burden already associated with behavioral weight loss sessions, it is important to identify strategies to increase access that are both feasible and acceptable in the target population. Currently the feasibility and acceptability of an online family dyadic skills training is unknown among Black adults.

TEAM+ is an in-person 3-month family enhanced BWL intervention designed for Black adults consisting of a family dyadic skills training and core behavioral weight loss sessions. For this proposed pilot study, 20 black adults interested in weight loss will be recruited with a family member committed to attending both the skills training and core sessions. Participants must 1) be ≥18 years of age, 2) self-identify as Black/African American, 3) reside in the Raleigh/Durham/Chapel Hill area, and 4) have internet access. The core sessions will be delivered in person. To test the feasibility and acceptability of an interactive counselor-led online training, the family dyadic skills training will be delivered online using a web-conferencing platform (e.g., Zoom).

ELIGIBILITY:
Inclusion Criteria:

* self-identify as a Black or African American,
* are between 18-75 years old
* have a family member willing to attend study session with you
* have Internet access
* reside in the Raleigh/Durham/Chapel Hill area,

Exclusion Criteria:

* not interested in losing weight
* have any conditions affecting weight
* currently receiving cancer treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Candice Alick, PhD, MS, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Center for Health Promotion and Disease Prevention, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved from an IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a dyad based study in which each Index Participant(IP) was invited to enroll with a Family Member(FM). In some cases, FM also chose to enroll as IP as part of the related dyad. The reported data reflect all enrolled IP, including those who were also FM. FM not enrolled as IP were nonetheless represented in the participant flow as FM. No data were collected for FM who did not enroll as IP. As such, these individuals are not represented in any of the reported data.
Period: Overall Study
Arm/Group | In-person Family Skills Training | Online Family Skills Training
Started | 11 | 10
Index Partners (Including Family Members Enrolled as Index Partners) | 11 | 8
Family Members (Non-Index Partners) | 0 | 2
Completed | 11 | 8
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Population: This study utilized a dyadic design, wherein each Index Participant (IP) was invited to enroll alongside a Family Member(FM). In certain cases, FM also elected to enroll as IP (together with an IP). The reported enrollment figures reflect all individuals who were formally enrolled as IP. No data were collected for FM who did not enroll as IP; therefore, these individuals are not represented in the reported data.
Groups:
- In-person Family Skills Training: The index partner participated in intervention as a dyad with a family member with an in-person skills training.
  Together, Eating and Activity, Matter Plus (TEAM+) In-Person: TEAM+ is a 3-month, family enhanced behavioral weight loss (BWL) intervention designed for Black adults consisting of in-person family dyadic skills training and core behavioral weight loss sessions.
- Online Family Skills Training: The index partner participated in intervention as a dyad with a family member with an online skills training.
  Together, Eating and Activity, Matter Plus (TEAM+) Online: TEAM+ is a 3-month, family enhanced behavioral weight loss (BWL) intervention designed for Black adults consisting of an online family dyadic skills training and in-person core behavioral weight loss sessions.
- Total: Total of all reporting groups
Arm/Group | In-person Family Skills Training | Online Family Skills Training | Total
Number analyzed (Participants) | 11 | 8 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.27 (13.76) | 54.13 (13.15) | 49.58 (14.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 5 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 8 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 8 | 19
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight
Description: Body weight (kg) expressed as a continuous variable will be collected on a digital scale.
Time Frame: Baseline, 12 weeks
Population: Overall Number of Participants Analyzed in this measure includes Index Participants. Family Member who were part of a dyad did not participate in data collection are not included in the reported numbers.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | In-person Family Skills Training | Online Family Skills Training
Number analyzed (Participants) | 11 | 8
kg | -0.91 (4.83) | -2.92 (4.04)

2. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Body mass index calculated from kg/m^2.
Time Frame: Baseline,12 weeks
Population: All collected data are reported. Two participants (one from the in-person) could not have their height recorded during the assessment. Overall Number of Participants Analyzed in this measure includes Index Participants. Family Member who were part of a dyad did not participate in data collection are not included in the reported numbers.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | In-person Family Skills Training | Online Family Skills Training
Number analyzed (Participants) | 9 | 8
kg/m^2 | -0.27 (2.05) | -0.77 (1.33)

3. Secondary Outcome: Change in Self-Regulation of Eating Behaviors
Description: The Eating Behavior Inventory (EBI) 20 items measures the adoption of eating behaviors associated with weight loss (e.g., monitoring quantity eaten, frequency of weighing, shopping from a list) to measure self-regulation behaviors. Items are rated on a 5-point frequency scale from "never or hardly ever" to "always or almost always." Scores range from 26 to 130. Items are scored such that higher scores indicate eating patterns that are considered more "appropriate" or facilitative of weight control.
Time Frame: Baseline,12 weeks
Population: All collected data are reported. Two participants (one from each Arm) did not complete the EBI. Overall Number of Participants Analyzed in this measure includes Index Participants. Family Member who were part of a dyad did not participate in data collection are not included in the reported numbers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In-person Family Skills Training | Online Family Skills Training
Number analyzed (Participants) | 10 | 7
score on a scale | 7.2 (11.21) | 9.29 (11.28)

4. Secondary Outcome: Change in Self-Efficacy of Eating Behaviors
Description: Measured by survey responses to the Weight Efficacy Lifestyle Questionnaire Short Form (WEL-SF).Scale goes from 0 (not at all confident) to 10 (very confident). Higher scores mean better self efficacy. The total score on the WEL-SF ranges from 0 to 80, with higher scores indicating greater self-efficacy in controlling eating behaviors. There are 8 items. This information presented here represents change scores from baseline to post intervention.
Time Frame: Baseline,12 weeks
Population: All collected data are reported. Three participants (two from the in-person arm and one from the online arm) did not complete the WEL-SF. Overall Number of Participants Analyzed in this measure includes Index Participants. Family Member who were part of a dyad did not participate in data collection are not included in the reported numbers.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In-person Family Skills Training | Online Family Skills Training
Number analyzed (Participants) | 9 | 7
units on a scale | 13.63 (18.02) | 9.43 (27.40)

5. Secondary Outcome: Change in Social Support Effectiveness
Description: Social Support Effectiveness Survey (25 items) measures partner social support effectiveness. The measure includes items assessing the quantity and quality (e.g., "To what extent did you wish this person's advice or information had been different somehow-for instance, a different type of help, or offered in a different way or at a different time?") on a rating scale ranging from "not at all" to "extremely" for 3 types of support (e.g., emotional, informational, and instrumental). The measure also assesses negative byproducts of support provided (e.g., feelings of guilt or indebtedness) using Yes/No options. All responses are numerically transformed. Total scores range from 0 to 80, with higher scores indicating more effective support.
Time Frame: Baseline,12 weeks
Population: All collected data are reported. Four participants (two from the in-person arm and two from the online arm) did not complete the Social Support Effectiveness Survey. Overall Number of Participants Analyzed in this measure includes Index Participants. Family Member who were part of a dyad did not participate in data collection are not included in the reported numbers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In-person Family Skills Training | Online Family Skills Training
Number analyzed (Participants) | 9 | 6
score on a scale | 2.67 (10.07) | -9.0 (6.14)

6. Secondary Outcome: Change in Social Support for Eating
Description: The Social Support and Eating Habits Survey (10 items) measures social support specific to healthy eating. Assess encouragement for eating behaviors from partners (e.g., "Encouraged me not to eat 'unhealthy food' when I am tempted") and discouragement for eating behaviors from partners (e.g., "Brought home foods I am trying not to eat"). The items are rated on a scale of "none" to "very often." Total scores range from 5 to 50, with higher scores indicating more social support for eating behaviors.
Time Frame: Baseline,12 weeks
Population: All collected data are reported. Two participants (two from the in-person arm and one from the online arm) did not complete the Social Support and Eating Habits Survey. Overall Number of Participants Analyzed in this measure includes Index Participants. Family Member who were part of a dyad did not participate in data collection are not included in the reported numbers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In-person Family Skills Training | Online Family Skills Training
Number analyzed (Participants) | 10 | 7
score on a scale | 24.1 (14.22) | 30.43 (13.80)

7. Secondary Outcome: Change in Social Support for Exercise
Description: The exercise participation subscale of the Social Support and Exercise Survey (10 items) measures social support specific to exercise behaviors assessing the level of support for exercise from partners. Subscale example items include "Exercised with me" and "Criticized or made fun of me for exercising." Total scores range from 5 to 50, with higher scores indicating more social support for exercise participation behaviors.
Time Frame: Baseline,12 weeks
Population: All collected data are reported. Three participants (one from the in-person arm and two from the online arm) did not complete the Social Support and Exercise Survey. Overall Number of Participants Analyzed in this measure includes Index Participants. Family Member who were part of a dyad did not participate in data collection are not included in the reported numbers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In-person Family Skills Training | Online Family Skills Training
Number analyzed (Participants) | 10 | 6
score on a scale | -0.8 (11.46) | 1.67 (9.53)

8. Secondary Outcome: Change in Family Communication
Description: Family communication is assessed with the communication subscale of the McMaster Family Assessment Device (6 items). Communication is defined as the exchange of information among family members. Items focused on whether verbal messages were clear and direct for the intended recipient. Responses ranged from "strongly agree" to "strongly disagree." . Uses a 4-point Likert scale for responses, ranging from "strongly disagree" to "strongly agree", subscale 1-4. Total score range 6-24. Higher scores represent unhealthy communication. Change score from baseline to post intervention presented here.
Time Frame: Baseline, 12 weeks
Population: All collected data are reported. Four participants (two from the in-person arm and two from the online arm) did not complete the McMaster Family Assessment Device Communication scale. Overall Number of Participants Analyzed in this measure includes Index Participants. Family Member who were part of a dyad did not participate in data collection are not included in the reported numbers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In-person Family Skills Training | Online Family Skills Training
Number analyzed (Participants) | 9 | 6
score on a scale | 0 (1.70) | 1.67 (3.86)

9. Secondary Outcome: Change in Family Cohesion
Description: The cohesion subscale (10 items) of the Family Adaptability and Cohesion Evaluation Scale III measures the emotional bonding family members have with one another. Items like "Family members ask each other for help" rated on a 5-point Likert scale from "almost never" to "almost always." The score has a range of 10 to 50.
Time Frame: Baseline, 12 weeks
Population: All collected data are reported. Four participants (two from the in-person arm and two from the online arm) did not complete the Family Adaptability and Cohesion Evaluation Scale III. Overall Number of Participants Analyzed in this measure includes Index Participants. Family Member who were part of a dyad did not participate in data collection are not included in the reported numbers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In-person Family Skills Training | Online Family Skills Training
Number analyzed (Participants) | 9 | 6
score on a scale | -0.67 (4.37) | 6 (7.92)

10. Secondary Outcome: Change in Family Emotional Involvement
Description: The family emotional involvement (7 items) of the Family Emotional Involvement and Criticism Scale rate items on a 5-point Likert scale. The scale has a range of 7 to 35. Higher scores on the emotional involvement subscale indicate higher levels of perceived emotional involvement.
Time Frame: Baseline, 12 weeks
Population: All collected data are reported. Four participants (two from the in-person arm and two from the online arm) did not complete the Family Emotional Involvement and Criticism Scale. Overall Number of Participants Analyzed in this measure includes Index Participants. Family Member who were part of a dyad did not participate in data collection are not included in the reported numbers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In-person Family Skills Training | Online Family Skills Training
Number analyzed (Participants) | 9 | 6
score on a scale | 0.22 (2.78) | 2.33 (3.09)

11. Secondary Outcome: Change in Family Perceived Criticism
Description: The perceived criticism (7 items) subscales of the Family Emotional Involvement and Criticism Scale rate items like on a 5-point Likert scale. The scale has a range of 7 to 35. Higher scores on the perceived criticism scale indicate higher levels of perceived emotional involvement.
Time Frame: Baseline, 12 weeks
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In-person Family Skills Training | Online Family Skills Training
Number analyzed (Participants) | 9 | 6
score on a scale | -1.67 (2.98) | -1.67 (4.11)

12. Secondary Outcome: Change in Family Collaborative Problem Solving
Description: The Family Problem-Solving Communication Index (10 items) was used to measure the specific communication style that families use to manage and solve problems and conflicts in various types of stressful situations. The 2 subscales are combined to report a total score for affirmatory communication and incendiary communication combined, the response options were "false," "mostly false," "mostly true," and "true." Scores range from 10 to 50 and a higher/lower score reflects a worse problem solving skills.
Time Frame: Baseline, 12 weeks
Population: All collected data are reported. Four participants (two from the in-person arm and two from the online arm) did not complete the Family Problem-Solving Communication Index. Overall Number of Participants Analyzed in this measure includes Index Participants. Family Member who were part of a dyad did not participate in data collection are not included in the reported numbers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In-person Family Skills Training | Online Family Skills Training
Number analyzed (Participants) | 9 | 6
score on a scale | -0.11 (3.03) | 0.67 (2.23)

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through study completion, a total of up to 3 months.
Description: Adverse Events data were collected for index partners and family members who chose to be participants at baseline and had outcome data collected. For family members who did not choose to participate in data collection as full participants, adverse events were not collected.
Groups:
- In-person Family Skills Training: The index partner will participate in intervention as a dyad with a family member with an in-person skills training.
  Together, Eating and Activity, Matter Plus (TEAM+) In-Person: TEAM+ is a 3-month, family enhanced behavioral weight loss (BWL) intervention designed for Black adults consisting of in-person family dyadic skills training and core behavioral weight loss sessions.
  Baseline data were not collected from family members
- Online Family Skills Training: The index partner will participate in intervention as a dyad with a family member with an online skills training.
  Together, Eating and Activity, Matter Plus (TEAM+) Online: TEAM+ is a 3-month, family enhanced behavioral weight loss (BWL) intervention designed for Black adults consisting of an online family dyadic skills training and in-person core behavioral weight loss sessions.
  Baseline data were not collected from family members.
Arm/Group | In-person Family Skills Training | Online Family Skills Training
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/8
Other Adverse Events (participants affected / at risk) | 0/11 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/08/NCT05981508/Prot_SAP_001.pdf
  • Informed Consent Form (2023-08-17): https://cdn.clinicaltrials.gov/large-docs/08/NCT05981508/ICF_000.pdf